CLINICAL TRIAL: NCT04843384
Title: The Effect of Reiki on Anxiety, Stress, and Comfort Levels Before Gastrointestinal Endoscopy
Brief Title: The Effect of Reiki on Anxiety, Stress, and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, HEDİYE UTLİ, PhD, RN, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hediye
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Reiki; Gastro-Intestinal Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki (Experimental): Experimental
  Interventions: Other: Reiki
- Sham reiki (Sham Comparator): Sham Comparator
  Interventions: Other: Sham reiki
- Control (No Intervention): Control

INTERVENTIONS:
Other: Reiki — Reiki
  Arms: Reiki
Other: Sham reiki — sham Reiki
  Arms: Sham reiki

SUMMARY:
Upper gastrointestinal (GI) endoscopy is a procedure that is used in the examination, diagnosis, and treatment of the esophagus, stomach, and duodenum. With developments in present-day technology, it is safe and widely used. This study's aim is to determine the effect of Reiki when applied before upper gastrointestinal endoscopy on levels of anxiety, stress, and comfort. This single-blind, randomized, sham-controlled study was held between February and July 2021.

DETAILED DESCRIPTION:
Anxiety and stress are problems that are often seen in patients undergoing upper GI endoscopy, and managing them is an important step in calming the patient and thereby reducing complications.The results of this study will contribute to the literature in forming a basis for other studies on the topic. The aim of this study is to evaluate the effects of the application of Reiki and sham Reiki on anxiety, stress, and comfort levels in patients undergoing upper GI endoscopy.

ELIGIBILITY:
Inclusion criteria

* patients who were having an upper GI endoscopy for the first time,
* patients who were age 18 or over,
* patients who had not previously had Reiki or sham Reiki (SR),
* patients who did not have a history of an operation in the previous six months,
* patients who were not using anxiolytic, hypnotic, or sedative drugs,
* patients who had no cognitive or effective problems or any hindrance in communication,
* patients who was literate, and who agreed to take part in the study.

Exclusion criteria

* patients who had an upper GI endoscopy with more than one elective condition,
* patients who was undergoing an emergency upper GI endoscopy,
* patients who were using anxiolytic, hypnotic, or sedative drugs,
* patients who had taken an opioid analgesic before the procedure,
* patients who completed the data collection forms incorrectly or incompletely,
* patients who had previously had Reiki or SR,
* patients who had a runny nose, fever, cough or any complaint of breathing difficulty,
* patients who were not literate and who did not wish to voluntarily participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Stress (VASS) | "Average of 1 year"
  The VASS reliably assesses levels of perceived stress.The VASS used in this study is a horizontal line with two points labeled "No stress" and "High stress" at a distance of 0 and 10 cm from each other.
State Anxiety Inventory (SAI) | "Average of 1 year"
  The SAI was developed by Spielberger et al., and the validity and reliability of the Turkish version were tested by Oner and Le Compte in 1974 to 1977.The highest possible score is 80, and the lowest is 20.
Short General Comfort Questionnaire (SGCQ) | "Average of 1 year"
  The SGCQ was devised by Kolcaba et al. in 2006 and adapted to Turkish society by Citlik et al. in 2018. It consists of 28 items, and the items on the scale score between 28 and 168 in total.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül VURAL DOĞRU, PhD, Study Chair — Mersin University
Locations (1):
- Hediye Utli, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No